CLINICAL TRIAL: NCT04022200
Title: Long Term Clinical Outcomes of Angioplasty With Paclitaxel-coated Balloon Only Strategy for Coronary de Novo Lesions: a Single Center Registry Study
Brief Title: Angioplasty With Paclitaxel-coated Balloon Only Strategy for Coronary de Novo Lesions
Acronym: DCB-denovo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Xue Yu, Vice Director of Cardiology Department, Beijing Hospital
Other Study IDs: BJH DCB for de novo
Record Dates: First submitted 2019-07-14; First posted 2019-07-17 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Coronary Disease
Keywords: drug-coated balloon; angioplasty; de novo lesions
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paclitaxel DCB for De Novo Coronary Lesions: we define de novo coronary artery lesions as the lesions never been treated with any interventional device, such as POBA, stent, rota ablation, laser etc.
  Interventions: Device: Paclitaxel DCB

INTERVENTIONS:
Device: Paclitaxel DCB — The length of the DCB catheter should be chosen to exceed the target lesion for at least 2mm (at both proximal and distalends). The catheter(s) will be inflated for 30 to 60s with a minimum of 7 atm. Predilation of the diseased coronary segment with a uncoated balloon/scoring balloon/cutting balloon before the use of DCB will be encouraged. DES should be implanted if the angiographic result after DCB alone therapy is not satisfactory due to significant recoil/residual stenosis or dissection (Type C-F).

SUMMARY:
Drug-coating balloon (DCB) is a new interventional device for treatment of obstructive coronary artery disease (CAD). There is limited data on the long term efficacy and safety of DCB-only strategy for coronary de novo lesions in Asian patients. We therefore carry out this registry study to evaluated the clinical outcomes of paclitaxel DCB in Chinese patients in a real world medical practice.

DETAILED DESCRIPTION:
DCB has emerged as a new interventional option to treat obstructive CAD. Characterized by non-stent-based local drug delivery system, DCB has several advantages over drug-eluting stent(DES).Paclitaxel DCB inhibits excessive neointimal hyperplasia of a diseased lesions without leaving a permanent metallic frame, therefore reducing the risk of coronary thrombosis and eliminating adverse events associated with stent fracture, allergic reactions to metal struts or polymer. Since only 1 to 3 months duration of dual anti-platelet therapy(DAPT) is required after DCB intervention, the bleeding risk associated with prolonged DAPT is reduced. DCB angioplasty was proved safe in an all-comers, prospective, multicenter registry and confirmed not inferior to DES when treating small coronary lesions in a randomized clinical trial(BASKET SMALL-2). DCB has been used in"off-label"indications in the"real world" for de novo lesions, especially in vessels with diameter more than 2.75mm, and there is limited data on its long term clinical efficacy and safety in Asian patients in contemporary clinical registries. We therefore sought to evaluate the long term clinical outcome of DCB in treatment of coronary de novo lesions in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient-related criteria：

   * Patients with stable angina, unstable angina, myocardial infarction or evidence of asymptomatic myocardial ischemia and consent to receive coronary intervention therapy;
   * Consent to receive clinical follow up at 30 days, 3, 6, 12 and 24 months.
   * Consent to receive one angiographic follow up at 24 months after procedure.
2. Lesion-related criteria：

   * Target coronary lesions without previous intervention therapy;
   * The lesions was intervened only with DCB;
   * The distance between other lesions requiring intervention therapy and the target lesion must >10mm.

Exclusion Criteria:

1. Patient-related criteria：

   * Severe congestive heart failure[LVEF <30% or NYHA( New York Heart Association) III/IV)]
   * Severe valvular heart disease;
   * Pregnant or breastfeeding women;
   * Life expectancy no more than 1 year or factors causing difficulties in clinical follow up;
   * Bleeding predisposition, contraindications of anticoagulants or antiplatelet agents;
   * Intorerance to aspirin and/or clopidogrel or other anti platelet drugs;
   * Leukopenia or thrombopenia;
   * Stroke within 6 months prior to the operation;
   * A history of severe hepatic or renal failure.
2. Lesion-related criteria ：

   * Ostia lesions of left main or right coronary artery;
   * Percutaneous coronary intervention of the graft vessel;
   * Lesions that are not indications of PTCA(percutaneous transluminal coronary angiography) or other intervention therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina, unstable angina, myocardial infarction or evidence of asymptomatic myocardial ischemia and consent to receive coronary intervention therapy. They will receive clinical follow up at 30 days, 3, 6, 12 and 24 months after procedure and one angiographic follow up at 24 months after procedure.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The rate of net adverse cardiac events (NACEs) at 24 months after DCB treatment. | Clinical follow-up at 24 months after the procedure.
  A composite endpoint of NACEs, including cardiovascular death, myocardial infarction, target lesion revascularization, target vessel revascularization, stroke, all cause bleeding.

SECONDARY OUTCOMES:
Late lumen loss(LLL) at 24 months follow-up | Coronary angiography follow-up at 24 months after the procedure.
  LLL is defined as minimal lumen diameter(MLD) at follow-up minus MLD immediately post the procedure according to QCA.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yu, MD, Study Chair — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu X, Ji F, Xu F, Zhang W, Wang X, Lu D, Yang C, Wang F. Treatment of large de novo coronary lesions with paclitaxel-coated balloon only: results from a Chinese institute. Clin Res Cardiol. 2019 Mar;108(3):234-243. doi: 10.1007/s00392-018-1346-8. Epub 2018 Aug 3. PMID 30074078
- [Background] Ann SH, Her AY, Singh GB, Okamura T, Koo BK, Shin ES. Serial Morphological and Functional Assessment of the Paclitaxel-coated Balloon for de Novo Lesions. Rev Esp Cardiol (Engl Ed). 2016 Nov;69(11):1026-1032. doi: 10.1016/j.rec.2016.03.026. Epub 2016 Jun 16. English, Spanish. PMID 27321644
- [Background] Nishiyama N, Komatsu T, Kuroyanagi T, Fujikake A, Komatsu S, Nakamura H, Yamada K, Nakahara S, Kobayashi S, Taguchi I. Clinical value of drug-coated balloon angioplasty for de novo lesions in patients with coronary artery disease. Int J Cardiol. 2016 Nov 1;222:113-118. doi: 10.1016/j.ijcard.2016.07.156. Epub 2016 Jul 27. PMID 27494722
- [Background] Shin ES, Ann SH, Balbir Singh G, Lim KH, Kleber FX, Koo BK. Fractional flow reserve-guided paclitaxel-coated balloon treatment for de novo coronary lesions. Catheter Cardiovasc Interv. 2016 Aug;88(2):193-200. doi: 10.1002/ccd.26257. Epub 2015 Oct 1. PMID 26423017